CLINICAL TRIAL: NCT02344732
Title: Effect of Systemic Oxygen on Corneal Epithelial Wound Healing in Diabetic Patients Undergoing Pars Plana Vitrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Teh Wee Min, Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMRR-13-449-15617
Record Dates: First submitted 2015-01-08; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Corneal Diseases
Keywords: epithelium, cornea, diabetes, vitrectomy, oxygen
MeSH Terms: conditions — Corneal Diseases; Diabetes Mellitus | interventions — Dexamethasone; Neomycin; Maxitrol; homatropine; nitrox

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Group (Active Comparator): topical Maxitrol™ six-hourly and homatropine 2% six-hourly
  Interventions: Drug: Dexamethasone 0.1%, Neomycin Sulfate and Polymyxin B Sulfate topical eye drops four times daily; Drug: Homatropine 2% eye drops thrice daily
- Oxygen Group (Experimental): standard medical treatment of topical Maxitrol™ six-hourly and homatropine 2% six-hourly, plus systemic oxygen via simple face mask at 10 litres/min for one hour, in 12-hourly sessions for 3 days
  Interventions: Drug: Dexamethasone 0.1%, Neomycin Sulfate and Polymyxin B Sulfate topical eye drops four times daily; Drug: Homatropine 2% eye drops thrice daily; Drug: Oxygen gas

INTERVENTIONS:
Drug: Dexamethasone 0.1%, Neomycin Sulfate and Polymyxin B Sulfate topical eye drops four times daily
  Other Names: Maxitrol
Drug: Homatropine 2% eye drops thrice daily
Drug: Oxygen gas
  Arms: Oxygen Group

SUMMARY:
1. To compare the corneal epithelial defect healing time between diabetic patients receiving and not receiving supplementary oxygen after vitrectomy.
2. To determine whether factors such as age, duration of diabetes, duration of surgery and level of glycemic control have any influence on corneal epithelial wound healing time in diabetic patients receiving and not receiving supplementary oxygen post-vitrectomy.

DETAILED DESCRIPTION:
This study aims to determine whether systemic oxygen therapy delivered through face mask would have beneficial effects on the healing of corneal epithelial wound in post-vitrectomy diabetic patients. It will be a prospective, randomised interventional clinical study conducted on diabetic patients indicated for vitrectomy. Rationale of this study is to see if systemic oxygen delivered via face mask will hasten the resolution of corneal epithelial defects, which may either be iatrogenic (surgically-induced intra-operatively to enable clearer visualisation for the surgeon) or spontaneous (due to corneal epithelial fragility which is commoner in diabetics)

ELIGIBILITY:
Inclusion Criteria:

* diabetic patients aged 18 years and above planned for pars plana vitrectomy that required intra-operative corneal epithelial debridement to allow better surgical visualisation of the fundus were recruited within the study duration

Exclusion Criteria:

* pre-existing ocular surface or corneal disease, recent eye surgery within one month from the vitrectomy, glaucoma and if the patients have any contraindications to oxygen therapy (e.g. chronic obstructive pulmonary disease).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Mean corneal epithelial wound healing time (in days) | 1 to 7 days

SECONDARY OUTCOMES:
Age of subject as a factor influencing wound healing time | 1-7 days
Glycemic control of subject (measured by glycated hemoglobin, HbA1c) | 1-7 days
Duration of surgery and its influence on wound healing time | 1-7 days
Duration of diabetes mellitus (measured in years) and its influence on wound healing time | 1-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Wee-Min Teh, MD, Principal Investigator — Universiti Sains Malaysia